CLINICAL TRIAL: NCT01378403
Title: Evaluation of Dorsal Visual Stream in Patients With Schizophrenia
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Revital Amiaz, MD - Senior Psychiatrist, Psychiatry clinic, Sheba Medical Center
Other Study IDs: SHEBA-07-4545-RA-CTIL
Record Dates: First submitted 2011-06-20; First posted 2011-06-22 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Cognitive deficites; Degraded objects; Magnocellular pathway
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Schizophrenia patients in comparing to normal controls show decreased ability to identify objects with decreased level of fragmentation, a task that is associated with magnocellular pathway function.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia

Exclusion Criteria:

* Ophthalomological or Neurological problems
* Left handed

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients suffering from schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2007-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Revital Amiaz, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Psychiatry Clinic - Sheba Medical Center, Ramat Gan, Israel